CLINICAL TRIAL: NCT04720352
Title: PURSUIT: Prospective US Radiofrequency SUI Trial
Brief Title: Prospective US Radiofrequency SUI Trial
Acronym: PURSUIT
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: Viveve Inc. (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: VI-17-06
Record Dates: First submitted 2021-01-18; First posted 2021-01-22 (Actual); Last update posted 2021-07-26 (Actual); Status verified 2021-07

CONDITIONS: Urinary Incontinence, Stress
MeSH Terms: conditions — Urinary Incontinence, Stress

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: Yes | Unapproved Device: Yes

ARMS (2):
- Sham Comparator (Sham Comparator): Sham delivers non therapeutic levels of radiofrequency and cryogen
  Interventions: Device: Sham
- Active Arm (Experimental): Active arm delivers radiofrequency and cryogen
  Interventions: Device: Active treatment

INTERVENTIONS:
Device: Active treatment — Active treatment delivers radiofrequency and cryogen
  Arms: Active Arm
Device: Sham — Sham delivers non therapeutic levels of radiofrequency and cryogen
  Arms: Sham Comparator

SUMMARY:
PURSUIT: Prospective US Radiofrequency SUI Trial (VI-17-06) is a prospective, randomized, sham controlled, double blind study in premenopausal women with stress urinary incontinence. The study will be conducted in 390 subjects, randomized 2:1 with active or sham treatment. Study duration is 12 months post treatment. The primary objective is to evaluate the efficacy of the Viveve treatment, SUI protocol, in improving mild to moderate stress urinary incontinence (SUI), assessed using the 1-hour Pad Weight Test for up to 12 months post-treatment.

DETAILED DESCRIPTION:
PURSUIT: Prospective US Radiofrequency SUI Trial (VI-17-06) is a prospective, randomized, sham controlled, double blind study in premenopausal women with stress urinary incontinence. The study will be conducted in 390 subjects, randomized 2:1 with active or sham treatment. Study duration is 12 months post treatment. The primary objective is to evaluate the efficacy of the Viveve treatment, SUI protocol, in improving mild to moderate stress urinary incontinence (SUI), assessed using the 1-hour Pad Weight Test for up to 12 months post-treatment. Secondary endpoints include:

* Percent of subjects who are responders in the 1-hour Pad Weight Test at 3- and 6-months post-treatment.
* Change from Baseline (CFB) to 3, 6- and 12-months post-treatment in the number of incontinence episodes as assessed by the 3-day bladder voiding diary.
* Percent of subjects with no incontinence episodes at 3, 6- and 12-months post-treatment as assessed by the 3-day bladder voiding diary.
* CFB to 3, 6, 9- and 12-months post-treatment in the I-QOL, ICIQ-UI-SF, PGI-I and MESA questionnaires.
* Percent CFB to 3, 6- and 12-months post-treatment in the 1-hour Pad Weight Test.

ELIGIBILITY:
Inclusion Criteria:

I.1 Able to understand and has voluntarily signed and dated the most current informed consent form (ICF) prior to initiation of any screening or study-specific procedures.

I.2 Willing to comply with study requirements and instructions.

I.3 Symptoms and diagnosis of stress urinary incontinence as determined by the following:

1. If there are mixed symptoms there must be a predominant stress component as determined by the 3-day diary results and MESA questionnaire
2. Patient-reported or history of SUI symptoms for > 6 months prior to screening.
3. Positive Bladder Stress Test at the Baseline Visit.
4. Positive Q-tip test at the Baseline Visit (the observation of an angle that exceeds 30 degrees from horizontal in the opinion of the investigator or designee to denote hypermobility).
5. 1-hour pad weight at the Baseline Visit with a >10 and <50 g net increase from the pre-test pad weight.
6. Subjects must complete 3 days in the 3-day voiding diary during 3 consecutive days in the 7 days prior to the Baseline Visit, and subjects must report a minimum of 1 incontinence episode per day or > 4 incontinence episodes over the 3 days as reported in the 3-day voiding diary.
7. For the Baseline 3-day diary, subjects must be compliant with recording events (i.e. void, leak or fluid intake) as determined through coordinator interview with the subject and review of voids and fluid intake reported in the diary compared to normal daily measurements.

I.4 Pre-menopausal females, ≥18 years of age. Premenopausal is defined as a woman who has had menstrual cycles over the previous 12 months or who is determined to be premenopausal by the PI or sub-investigator (e.g. premenopausal woman with hysterectomy).

I.5 Body mass index (BMI) of ≤35 kg/m² at the Screening Visit. I.6 Normal, or abnormal but not clinically significant (i.e., mild atrophy with rugae present, low grade prolapse), physical, pelvic and neurologic exam at the Baseline Visit as determined by the investigator.

I.7 Negative urine pregnancy test at the Baseline and Randomization Visits and subject agrees to not become pregnant during the study and uses an acceptable form of birth control started at least 3 months prior to screening (with the exception of double barrier contraception, where the 3-months required prior to screening does not apply).

1. Examples of acceptable forms of birth control include: abstinence from heterosexual vaginal intercourse, hysterectomy, bilateral tubal ligation, vasectomy, double barrier contraception (note that condom and spermicide is not considered double barrier contraception), intrauterine device or hormonal contraceptive.
2. Rhythm and withdrawal are not considered acceptable forms of contraception.

Exclusion Criteria:

E.1 Currently breastfeeding or have discontinued breastfeeding fewer than 6 months prior to screening.

E.2 Undergone other stress urinary incontinence treatment(s), excluding behavioral modifications started >3 months prior to screening (e.g., Kegel exercises).

E.3 A MESA score of greater than 5 in sum on questions 10 - 12, or greater than 9 in sum on questions 10 - 15 at the screening visit (see appendix).

E.4 A post void residual measurement of greater than 150 ml as measured with ultrasound or bladder scanner at the screening visit.

E.5 Greater than 10 voids per day on average as measured with the 3-day diary at Baseline Visit.

E.6 Greater than 1 nocturia episode per day on average as measured with the 3-day diary at Baseline Visit.

E.7 Abnormal, clinically significant laboratory results at the Baseline Visit (as determined by the Investigator) that could impact the subject participation or evaluation for SUI. Retest is allowed with Sponsor approval.

E.8 Greater than 100 ounces of fluid consumed per day on average as measured with the 3-day diary at baseline Visit.

E.9 History of, or any current condition, illness, or surgery that might confound the results of urinary incontinence assessment, including, but not limited to:

1. Prominent (i.e., greater than Stage II pelvic organ prolapse as determined by a POP-Q evaluation (at Baseline) e.g., cystocele, rectocele
2. Neurological disorders (e.g., multiple sclerosis, Parkinson's disease, fibromyalgia)
3. Recurrent Urinary Tract Infections (UTI)
4. Current Urinary Tract Infection (UTI) as assessed by urine dipstick and associated urinary tract infection symptoms at the Baseline or Randomization Visit. If the subject has a UTI at the Baseline or Randomization Visit they may be treated with antibiotics, at the Investigator's discretion, and return within 7 days after UTI treatment completion.
5. Vesicoureteral reflux
6. Bladder stones
7. Bladder tumors
8. Interstitial cystitis E.10 Has any implantable electrical device [e.g., implantable pacemaker, automatic implantable cardioverter-defibrillator (AICD)].

E.11 A rectovaginal septum <2 cm. E.12 Planning on future pregnancies after the Viveve procedure.

E.13 Medical or immunological condition, including, but not limited to:

1. Uncontrolled cardiovascular, respiratory, neoplastic, infectious, and/or endocrinological condition that could impact the subject's ability to complete the trial.
2. Uncontrolled diabetes defined as hemoglobin A1c > 7%
3. Untreated chronic abdominal/pelvic pain disorder [including, but not limited to, dyspareunia, vaginismus, endometriosis, significant vulvovaginal atrophy (VVA), genitourinary syndrome of menopause (GSM), irritable bowel syndrome, or Crohn's disease].
4. Untreated medical condition or medication that, in investigator's opinion, may interfere with adequate wound healing response (e.g., congenital connective tissue disease) or the subject's ability to complete the clinical trial requirements.
5. Untreated active malignancy (with the exception of basal cell carcinoma of the skin) or undergoing treatment (using chemotherapeutic agents, radiation therapy, and/or cytostatic medications) that may interfere with adequate wound healing response or the subject's ability to complete the trial.
6. Untreated acute or chronic vaginal or vulvar disorder including, but not limited to, vulvovaginal atrophy/GSM; pain, including provoked/generalized vulvodynia, vulvar vestibulitis, dysesthetic vulvodynia, or vulvar dystrophy; current/chronic papulosquamous vulvar dermatoses (e.g., psoriasis, lichen planus, tinea cruris, lichen sclerosis, seborrheic dermatitis, contact/irritant dermatitis, lichen simplex, eczema); bullous dermatoses; systemic diseases with potential involvement of vulva; genital warts; past/current vaginal or vulvar radiotherapy or brachytherapy.
7. Active genital/pelvic infection (e.g., herpes, gonorrhea, chlamydia) observed on physical or pelvic exam at Baseline.
8. Active yeast infection. If the subject has an active vaginal yeast infection at the Baseline or Randomization Visit, they may be treated with an antifungal, at the Investigator's discretion, and return within 7 days after completion of vaginal yeast infection treatment.

E.14 Chronic use of anti-inflammatory drugs, including ibuprofen, aspirin, and oral steroids (excluding aspirin that is taken for cardiovascular prophylaxis).

E.15 Started taking any new medication, including herbal supplements and those taken in teas that potentially affects urination within 28 days prior to the Screening Visit, or had a change in the dosage of any medication that potentially affects urination within 28 days of the Screening Visit. Dosage should not change for the remainder of the study unless medically necessary.

E.16 Started or changed dose of local vaginal hormones <6 weeks before screening.

E.17 Undergone previous elective surgical or non-invasive procedure(s) in the vaginal canal (including previous treatment with the Viveve System or any other genital radiofrequency treatment; injectable bulking agent, cosmetic, laser, surgical, and/or genital enhancement procedure).

E.18 Participated in another clinical study within 6 months of screening or is not willing to abstain from participating in other clinical studies for duration of trial.

E.19 Employed by Viveve or participating investigative sites.

Min Age: 18 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 390 (Estimated)
Dates: Start 2021-01-11 (Actual); Primary Completion 2022-12-30 (Estimated); Study Completion 2022-12-30 (Estimated)

PRIMARY OUTCOMES:
1-hour pad weight test | 12 months
  Standard test of incontinence

SECONDARY OUTCOMES:
3-day diary | 3, 6, and 12 months
  Voiding diary
1-hour pad weight test | 3 and 6 months
  Standard test of incontinence
Patient Global Impression of Improvement (PGI-I) | 3, 6, 9, and 12 months
  Single question patient assessment
Medical, Epidemiologic, and Social aspects of Aging (MESA) questionnaire | 3, 6, 9, and 12 months
  Questionnaire for stress and urge incontinence
International Consultation on Incontinence Modular Questionnaire-Urinary Incontinence Short Form (ICIQ-UI-SF) | 3, 6, 9, and 12 months
  Incontinence severity, frequency QOL questionnaire
Incontinence Quality of Life (I-QOL) | 3, 6, 9, and 12 months
  QOL assessment

CONTACTS AND LOCATIONS:
Overall Officials: Eric S Rovner, MD, Principal Investigator — Medical University of South Carolina; Roger R Dmochowski, MD, Study Director — Vanderbilt University Medical Center
Locations (29):
- United States (29):
  - Coastal Clinical Research, Mobile, Alabama
  - Urological Associates of Southern Arizona, PC, Tucson, Arizona
  - Long Beach Clinical Trials Services, Inc., Long Beach, California
  - Emerson Clinical Research Institute, Washington D.C., District of Columbia
  - IntimMedicine Specialists, Washington D.C., District of Columbia
  - Multi-Specialty Research Associates, Inc, Lake City, Florida
  - A Premier Medical Research of Florida, Orange City, Florida
  - Florida Urology Partners, Tampa, Florida
  - Leavitt Clinical Research, Idaho Falls, Idaho
  - Cypress Medical Research Center, LLC, Wichita, Kansas
  - Research Integrity, LLC, Owensboro, Kentucky
  - Regional Urology, LLC, Shreveport, Louisiana
  - Chesapeake Urology Research Associates, Owings Mills, Maryland
  - Minnesota Women's Care, P.A., Maplewood, Minnesota
  - Boeson Research, Missoula, Montana
  - Adult and Pediatric Urology, Omaha, Nebraska
  - AccuMed Research Associates, Garden City, New York
  - Circuit Clinical, West Seneca, New York
  - Unified Women's Health Care of Raleigh, Raleigh, North Carolina
  - UWCR-Lyndhurst Clinical Research, Winston-Salem, North Carolina
  - Clinical Research Solutions, Middleburg Heights, Ohio
  - The Clinical Trial Center, LLC, Jenkintown, Pennsylvania
  - Hospital of the University of Pennsylvania, Philadelphia, Pennsylvania
  - Venus Gynecology, LLC, Myrtle Beach, South Carolina
  - Advances In Health Research, Houston, Texas
  - Cedar Health Research, Irving, Texas
  - Maximos OB/GYN, League City, Texas
  - Urology San Antonio, San Antonio, Texas
  - Health Research of Hampton Roads, Inc, Newport News, Virginia

IPD SHARING:
Plan to Share IPD: No